CLINICAL TRIAL: NCT06560619
Title: Tele-wellness Program for People With Disabilities: Mindfulness, Exercise, and Nutrition To Optimize Resilience (MENTOR)
Brief Title: Mindfulness, Exercise, and Nutrition To Optimize Resilience (MENTOR)
Acronym: MENTOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Wing Wong, Assistant Director, Center for Rehabilitation Outcomes Research, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00221578
Record Dates: First submitted 2024-08-14; First posted 2024-08-19 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Disabled Persons
Keywords: Mobility impairment; People with physical disability; Mindfulness; Exercise; Nutrition; Technology; Mobile health
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MENTOR Wellness Program (Experimental): MENTOR is an 8-week group program conducted via videoconferencing, designed for individuals with physical disabilities in the United States to enhance their health and well-being. The program includes 1 hour per week of mindfulness training, 2 hours per week of exercise, and 1 hour per week of nutrition education. Participants will also receive personalized health coaching and have access to a fitness instructor, registered dietician, and mindfulness coach. Additionally, participants will receive information on 8 other areas, including self-care skills, core values, outdoor time in nature, rest/relaxation, contributing to others, arts and leisure, relationships, and spiritual practice, all taught by a trained health coach over the 8-week period.
  Interventions: Behavioral: MENTOR

INTERVENTIONS:
Behavioral: MENTOR — Participants will attend a group-based, 8-week online program (a total of 40 hours) via Zoom videoconferencing. The program is split into three wellness sections (Mindfulness, Exercise, and Nutrition) and eight other sections (self-care skills, core values, outdoor time in nature, rest/relaxation, contribution to others, arts and leisure, relationships, and spiritual practice). Participants will access all assessment and intervention tools on any mobile device (phone, tablet, laptop, desktop) using a password-protected identification (ID) to log in via their devices. Health coaches can create intake flows to collect health data and track analytics. Participants can see their goals, upcoming intervention sessions, and activities through the study application (app). Features of the study app include goal setting, where participants record their goals, zoom videoconferencing links for online classes and coaching sessions, and the ability to share materials with participants.

SUMMARY:
The Mindfulness, Nutrition and Exercise to Optimize Resilience (MENTOR) program is offered through the National Center on Health, Physical Activity and Disability (NCHPAD). NCHPAD is funded by the Centers for Disease Control and Prevention (CDC), is a public health practice that offers health promotion programs and resources to people with mobility disabilities. The purpose of this project is to provide a free-of-charge wellness program designed to improve health and wellness for people with mobility and physical disability living in the United States.

DETAILED DESCRIPTION:
The objective of the MENTOR program is to improve wellness for people with mobility limitations. MENTOR is a free, 8-week program focusing on physical, mental, and emotional health for individuals with an existing disability or a recent diagnosis. The program provides core information on mindfulness, exercise, and nutrition. Participants get one-on-one health coaching and access to a fitness instructor, registered dietician, and mindfulness coach. The classes are virtual, and the exercise equipment needed for the classes will be mailed to participants.

The research question is to measure the effectiveness and implementation of the MENTOR program.

Participants will be asked to fill out an eligibility sign-up form on NCHPAD. If eligible, they will be consented by Shirley Ryan AbilityLab (SRAlab) via REDCap. On the same SRAlab REDCap survey link, after the consent form, they will be able to complete an interest form. If selected, participants will be asked to complete 3 surveys through NCHPAD Connect before the MENTOR program begins.

Once the 8-week MENTOR program is complete, you will be asked to complete a post-program survey for NCHPAD about your experience, and a post-program implementation survey through SRAlab.

ELIGIBILITY:
Inclusion Criteria:

* Lives in the United States
* People 18 years or older
* A self-reported physical disability/mobility limitation (or use an assistive device such as an ankle foot orthosis, cane, walker, scooter, or wheelchair).
* Have internet access and a mobile device (phone, tablet, laptop, desktop) to attend sessions.

Exclusion Criteria:

* Younger than 18 years old
* Living outside of the United States
* No physical disability/mobility limitation
* No internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Connor-Davidson Resilience Scale (CD-RISC) | Pre/Post 8-week Program
  This is a resilience measure to gain a better understanding of whether the program had any benefit to improving resilience. It consists of 10 items.The response scale has a 5-point range from 0 to 4. Scores are summed to provide a total score of 40, where higher scores indicate higher resilience. It measures the Effectiveness of the RE-AIM framework.

SECONDARY OUTCOMES:
Godin Leisure-Time Exercise Questionnaire (GLTEQ) | Pre/Post 8-week Program
  A self-report measure of physical activity. It is a 7-day recall questionnaire that contains 3 questions pertaining to light, moderate, and vigorous intensity activity. The GLTEQ can be scored either by summing all 3 intensity types (Total Activity score) after multiplying each by 3, 5, and 9, respectively, or by summing moderate and vigorous activity only (Health Promotion score). It measures the Effectiveness of the RE-AIM framework.
Mindfulness Attention Awareness Scale (MAAS) | Pre/Post 8-week Program
  This is a mindfulness scale which is used to identify potential changes in mindfulness.
  This scale contains 15 items that ask participants how frequently they have a certain experience, using a 6-point Likert scale from 1 to 6. The score is calculated by calculating the mean of these 15 items. Higher scores reflect more mindfulness. It measures the Effectiveness of the RE-AIM framework.
NCHPAD Wellness Assessment (NWA) | Pre/Post 8-week Program
  This assessment has 3 dimensions which are physical, mental, and emotional/spiritual health. Each dimension has 5 questions, and an additional question assesses the overall wellness (16 questions total). The NWA is scored on a Likert scale from 1-5. Higher scores reflect better wellness. It measures the Effectiveness of the RE-AIM framework.
Nutrition Questionnaire on Mindful Eating, Habits, and Knowledge | Pre/Post 8-week Program
  It is a survey to identify which dietary advice people find confusing. It consists of 3 domains: nutrition knowledge (24 items), mindful eating assessment (2 items), and eating habits (13 items).It measures the Effectiveness of the RE-AIM framework.
Global Health | Pre/Post 8-week Program
  It is a Patient-Reported Outcome Measurement Information System (PROMIS) Global Health Scale V1.2 for an overall evaluation of one's physical and mental health. It consists of 10 items. Raw scores can be converted to T-scores, with higher scores reflect better health. It measures the Effectiveness of the RE-AIM framework.

OTHER OUTCOMES:
Proportion of individuals who express interest in MENTOR | Pre Program (Week 1)
  This measure will be a proportion of contacted individuals who complete an eligibility survey. The proportion ranges from 0 to 100 percent. Higher percentages represent a higher reach. It measures the Reach domain in the RE-AIM framework.
Representativeness of individuals who express interest in MENTOR | Pre Program (Week 1)
  The sociodemographic and medical characteristics of individuals will be reviewed. It measures the Reach domain in the RE-AIM framework.
Proportion of eligible participants who begin MENTOR | Post Program (Week 8)
  This will measure the proportion of eligible participants who consent, complete a baseline survey, and start MENTOR. The proportion ranges from 0 to 100 percent. Higher percents represent a higher adoption. It measures the Adoption component of the RE-AIM framework.
Proportion of eligible participants who complete MENTOR | Post Program (Week 8)
  This will measure the proportion of eligible participants who retain and complete MENTOR. The proportion ranges from 0 to 100 percent. Higher percents represent a higher adoption. It measures the Adoption component of the RE-AIM framework.
Acceptability of Intervention Measure (AIM) | Post Program (Week 8)
  It measures the intervention's acceptability. This is a 4-item, 5-point Likert scale. Higher scores reflect higher acceptability. It measures the Implementation domain of the RE-AIM framework.
Intervention Appropriateness Measure (IAM) | Post Program (Week 8)
  It measures if the intervention is appropriate for intended users. This is a 4-item, 5-point Likert scale.Higher scores reflect higher appropriateness. It measures the Implementation domain of the RE-AIM framework.
Feasibility of Intervention Measure (FIM) | Post Program (Week 8)
  It measures if the intervention is feasible for use, dissemination, and delivery. This is a 4-item, 5-point Likert scale. Higher scores reflect higher feasibility. It measures the Implementation domain of the RE-AIM framework.
The likelihood of continuing the use of MENTOR | Post Program (Week 8)
  It will be measured by a single question: How likely are you to continue using MENTOR? It will be rated from 1-10 scale. Higher ratings represent a higher likelihood of continuing. It measures the Maintenance domain of the RE-AIM.
The likelihood of recommending MENTOR | Post Program (Week 8)
  It will be measured by a single question: How likely are you to recommend MENTOR to others? It will be rated from 1-10 scale. Higher ratings represent a higher likelihood of recommending. It measures the Maintenance domain of the RE-AIM.
Degree of difficulty to continue MENTOR for 6 months | Post Program (Week 8)
  It will be measured by a single question: How difficult are you to continue MENTOR for 6 months? It will be rated from the response options: extremely easy, moderately easy, slightly easy, neither easy nor difficult, slightly difficult, moderately difficult, extremely difficult. Participants choosing "extremely easy", "moderately easy", and "slightly easy" represent lower degree of difficulty, reflecting a higher maintenance. It measures the Maintenance domain of the RE-AIM.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Wong, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan Ability Lab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No